CLINICAL TRIAL: NCT06653439
Title: Analgesic Effect of Ultrasound-Guided Bilateral Subcostal Anterior Quadratus Lumborum Block in Laparoscopic Colorectal Surgery: A Randomized Controlled Trial
Brief Title: Analgesic Effect of Bilateral Subcostal Quadratus Lumborum Block in Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra Turunc, Assistant professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SQLB3CRS
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia; Regional Anesthesia; Post Operative Pain
Keywords: Anesthesia; Nerve block; Colorectal surgery; Subcostal Anterior Quadratus Lumborum Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Intervention Model Description: A block randomization was performed by an independent physician using a computer-generated sequence via a web-based program.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Researchers, surgeons and nurses, and those involved in study outcome analysis will not be aware of the randomization of the group. Due to the nature of the intervention, patient blinding was not feasible. Block quality and standardization will be performed by an anesthetist experienced in regional anesthesia for S-QLB block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S-QLB (Active Comparator): A bilateral S-QLB (20 ml, %0.25 bupivacaine, bilaterally) + IV morphine patient-controlled analgesia (PCA)
  Interventions: Procedure: Bilateral ultrasound guided Subcostal Quadratus Lumborum Block; Drug: IV morphine PCA
- Group Control (Active Comparator): IV morphine PCA
  Interventions: Procedure: Control; Drug: IV morphine PCA

INTERVENTIONS:
Procedure: Bilateral ultrasound guided Subcostal Quadratus Lumborum Block — Bilateral ultrasound-guided subcostal quadratus lumborum block (20 mL, 0.25% bupivacaine, bilaterally) will be performed. All patients will receive multimodal analgesia, including a single dose of IV tenoxicam 20 mg. Additionally, 15 mg/kg IV paracetamol (based on IBW) will be administered at skin closure and continued every 6 hours postoperatively. A standardized IV PCA protocol will be initiated using a PCA device programmed to deliver morphine boluses of 0.01-0.015 mg/kg (IBW), with a 6-minute lockout and a 4-hour maximum of 0.1-0.15 mg/kg (IBW). Upon arrival in the PACU, patients with a resting NRS ≥4 will receive titrated IV morphine boluses of 0.03 mg/kg (IBW; max 10 mg) every 10 minutes until pain is controlled. In the surgical ward, patients with breakthrough pain (NRS ≥4) despite PCA use will receive IV tramadol 1-1.5 mg/kg (IBW) in 50-100 mg slow doses, not exceeding 400 mg/day.All patients will receive 8 mg dexamethasone and 0.15 mg/kg ondansetron (IBW) for PONV prophylaxis.
  Other Names: S-QLB group
  Arms: Group S-QLB
Procedure: Control — Patients in this group will not undergo plane blocks. IV morphine PCA multimodal analgesia will be provided: all patients will receive a single dose of IV tenoxicam 20 mg. Additionally, 15 mg/kg IV paracetamol (based on IBW) will be administered at skin closure and continued every 6 hours postoperatively. A standardized IV PCA protocol will be initiated for all patients using a PCA device, programmed to deliver morphine boluses of 0.01-0.015 mg/kg (IBW), with a 6-minute lockout and a 4-hour maximum dose of 0.1-0.15 mg/kg (IBW). Upon arrival in PACU, patients with a resting NRS ≥4 will receive titrated IV morphine boluses of 0.03 mg/kg (IBW; max 10 mg) every 10 minutes until pain is controlled. In the ward, patients with breakthrough pain (NRS ≥4) despite PCA use will receive IV tramadol 1-1.5 mg/kg (IBW), administered slowly in 50-100 mg doses (max 400 mg/day). All patients will receive IV dexamethasone (8 mg) before induction and IV ondansetron (0.15 mg/kg IBW) near surgery end.
  Other Names: Control group
  Arms: Group Control
Drug: IV morphine PCA — A standardized IV PCA protocol will be initiated for all patients using a PCA device (Body Guard 575 pain manager, UK), programmed to deliver morphine boluses of 0.01-0.015 mg/kg (IBW), with a 6-minute lockout and a 4-hour maximum dose of 0.1-0.15 mg/kg (IBW). No basal infusion will be used.
  Other Names: PCA

SUMMARY:
Effective postoperative pain management is crucial for promoting early recovery and ambulation following laparoscopic colorectal surgery. Regional anesthesia techniques, like interfascial plane blocks, are increasingly being used to achieve this. The quadratus lumborum block (QLB) is a relatively new approach in abdominal surgeries, providing significant pain relief by blocking both somatic and sympathetic nerves. In particular, the anterior QLB technique allows local anesthetic to spread to the thoracic paravertebral space, making it potentially more effective for postoperative analgesia. The hypothesis of this study is that bilateral subcostal anterior QLB can reduce both postoperative pain and opioid consumption in laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
Postoperative pain management is a critical factor in enhancing recovery and ambulation following laparoscopic colorectal surgery. Effective analgesia is necessary to reduce complications, improve patient comfort, and shorten hospital stays. In this context, multimodal analgesia is a commonly used strategy that combines various analgesic drugs, such as paracetamol, nonsteroidal anti-inflammatory drugs (NSAIDs), and opioids, to manage pain more effectively by targeting different pathways.

Although opioids are considered the gold standard for postoperative pain control, their use is associated with several undesirable side effects, including nausea, vomiting, dizziness, constipation, and respiratory depression. These opioid-related complications can delay recovery, increase patient discomfort, and extend hospital stays. Therefore, minimizing opioid consumption while still providing effective pain relief is a primary goal in postoperative pain management, particularly for surgeries such as laparoscopic colorectal procedures.

To achieve this goal, regional anesthesia techniques have gained increasing popularity. These techniques, such as interfascial plane blocks, have the potential to reduce opioid use and improve pain control by targeting specific nerve pathways. One of the more recent approaches is the quadratus lumborum block (QLB), which involves the injection of local anesthetics near the quadratus lumborum muscle. This block is particularly useful in abdominal surgeries because it can provide pain relief by affecting both somatic and sympathetic nerves, leading to broader and more effective pain coverage.

The QLB has four different approaches: anterior, lateral, posterior, and intramuscular. The anterior QLB is of particular interest in this setting because it involves the injection of local anesthetic between the quadratus lumborum and psoas muscles, potentially allowing the anesthetic to spread into the thoracic paravertebral space. This spread could result in the blockade of both the somatic nerves and the thoracic sympathetic chain, offering more comprehensive pain relief that is beneficial for abdominal surgeries like colorectal procedures.

The potential advantages of the anterior QLB in laparoscopic colorectal surgery include reduced postoperative pain, decreased opioid consumption, and fewer opioid-related side effects. Additionally, regional anesthesia techniques like QLB may reduce postoperative complications, including respiratory issues, which are particularly important in abdominal surgeries that involve the diaphragm and lower thoracic nerves.

In this study, the hypothesis is that bilateral subcostal anterior QLB, administered during laparoscopic colorectal surgery, will significantly reduce both postoperative pain and the need for opioids.

The aim of this study is to investigate the effects of Bilateral subcostal anterior QLB on postoperative acute pain scores (0-24 hours) and 24- hour opioid consumption in patients who underwent laparoscopic colorectal surgery. Our study, which the investigators think will contribute to the literature, was planned as a prospective, randomized, controlled, parallel-group study.

Patients will be divided into two groups:

Group S-QLB:

A bilateral S-QLB (20 ml 0.25% bupivacaine + 1:400.000 adrenaline, bilaterally) will be performed. In addition, IV morphine-PCA will be applied postoperatively for 24 hours.

Group Control :

IV morphine-PCA will be applied postoperatively for 24 hours.

ELIGIBILITY:
Inclusion Criteria They will be aged between 18 and 75 years. They will have an American Society of Anesthesiologists (ASA) physical status classification of I to III.

They will be able to provide written informed consent.

Exclusion Criteria They will refuse to participate. They will have a body mass index (BMI) greater than 35 kg/m². They will have contraindications to peripheral nerve blocks (e.g., coagulopathy, abnormal INR, thrombocytopenia, local or systemic infection).

They will have clinically significant cardiovascular or cerebrovascular disease.

They will have severe hepatic, renal, or respiratory dysfunction. They will have known drug allergies. They will have a history of substance abuse. They will have chronic opioid use, defined as regular use of ≥15 mg oral morphine equivalent per day for at least 30 consecutive days within the past 3 months.

They will have chronic pain syndromes (e.g., fibromyalgia, diabetic neuropathy, or chronic low back pain).

They will have neuropsychiatric disorders or cognitive impairment that precludes effective communication with the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption in the first 24 hours after surgery | Postoperative day 1
  The primary outcome will be defined as cumulative opioid consumption during the first 24 hours following surgery, which will be calculated in intravenous morphine milligram equivalents (IV-MME), encompassing both PCA-administered morphine and rescue intravenous tramadol, according to the standardized ESAIC conversion guidelines. Patients can request opioids via a PCA device when their NRS score is≥ 4.

SECONDARY OUTCOMES:
Cumulative opioid consumption in the first 12 hours after surgery | Postoperative 12 hours.
  The secondary outcome will be defined as cumulative opioid consumption during the first 12 hours following surgery, calculated in intravenous morphine milligram equivalents (IV-MME). This will include both PCA-administered morphine and rescue intravenous tramadol, in accordance with the standardized ESAIC conversion guidelines. Patients may request opioids using a PCA device when their NRS score is ≥ 4.
Intraoperative Remifentanil Consumption | The remifentanil consumption will be recorded from anesthesia induction until the patient is referred to the recovery unit, up to 150 minutes.
  Total intraoperative remifentanil consumption will be recorded in micrograms (µg) from the start of anesthesia induction until the end of surgery.
Numerical Rating Scale Assessment of Postoperative Pain | Postoperative day 1
  Pain scores will be assessed using the 11-point Numerical Rating Scale (NRS), where 0 indicates no pain and 10 represents the worst imaginable pain. Evaluations will be performed both at rest (static) and during coughing or deep breathing (dynamic). Assessments will be conducted in the post-anesthesia care unit (PACU) after extubation and once communication is established, and subsequently at 3, 6, 12, 18, and 24 hours postoperatively.
Time to First Opioid Demand via PCA | Postoperative day 1
  Defined as the time elapsed from the patient's arrival in the post-anesthesia care unit (PACU) to the first patient-initiated opioid request via the patient-controlled analgesia (PCA) device.
Extent of Sensory Block | From block administration to 30 minutes post-procedure.
  Sensory block success was evaluated using a 3-point scale via pinprick testing of dermatomes T7 to L1 every 5 minutes after block administration. A successful block was defined as a sensory score ≥1. In all patients, a final dermatomal assessment was performed at the 30th minute to confirm block effectiveness, and the extent of dermatomal spread was documented.
The number of patients who required rescue analgesia. | Postoperative day 1
  The number of patients who required additional IV tramadol due to breakthrough pain (NRS ≥4) despite PCA use.
The patient number of Rescue antiemetic Requirement | Postoperative day 1
  All patients received standard prophylaxis for postoperative nausea and vomiting (PONV), including 8 mg IV dexamethasone before induction and 0.15 mg/kg IV ondansetron (based on ideal body weight) approximately 20 minutes before the end of surgery. PONV was assessed at 0, 3, 6, 12, 18, and 24 hours after extubation using a 5-point scale (0 = no nausea to 4 = multiple episodes of vomiting). Patients with a PONV score ≥3 received rescue treatment with 10 mg IV metoclopramide in 100 mL normal saline via slow infusion. The number of patients requiring rescue antiemetic therapy was recorded.
The number of patients with complications | Postoperative 7 days on an average
  The number of patients has any complications -directly related to the block or the drug used in the block- will be recorded
Mean Arterial Pressure | Postoperative day 1
  Intraoperative mean arterial pressure (MAP) values were recorded at predefined intervals to assess hemodynamic stability.
Heart Rate | Postoperative day 1
  Intraoperative heart rate values were recorded at predefined intervals to assess hemodynamic stability.
Time to First Mobilization | Postoperative day 3
  Defined as the time (in hours) from the end of surgery until the patient is first able to stand and ambulate postoperatively.
Time to First Flatus | Postoperative day 3
  Defined as the time (in hours) from the end of surgery to the first passage of flatus, serving as a clinical marker of return of bowel function.
Time to First Oral Intake | Postoperative day 3
  Defined as the time (in hours) from the end of surgery until the initiation of postoperative oral nutrition.
Length of Hospital Stay | Postoperative day 10
  Defined as the total postoperative hospital stay, measured in days, from the end of surgery until the patient meets institutional discharge criteria and is discharged from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Turunc, Study Director — Ondokuz Mayis University, School of Medicine, Department of Anesthesiology
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turunc E, Dost B, Kaya C, Ustun YB, Bilgin S, Ozdemir E, Koksal E, De Cassai A, Elsharkawy H. Efficacy of anterior subcostal quadratus lumborum block for postoperative analgesia in laparoscopic colorectal surgery: a randomized controlled trial. Reg Anesth Pain Med. 2025 Oct 28:rapm-2025-107136. doi: 10.1136/rapm-2025-107136. Online ahead of print. PMID 41151981